CLINICAL TRIAL: NCT00873561
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel, Dose-Ranging Study to Evaluate The Efficacy, Safety, Tolerability, and Pharmacodynamics of NBI-6024 In Adult and Adolescent Patients With New Onset Type 1 Diabetes Mellitus
Brief Title: A Study to Evaluate NBI-6024 in Adult and Adolescent Patients With New Onset of Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Chris O'Brien, Chief Medical Office and VP of Clinical Development, Neurocrine Biosciences Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NBI 6024-0101
Record Dates: First submitted 2009-03-27; First posted 2009-04-01 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes; type 1; adult; adolescent; new onset
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — NBI6024

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 Experimental (Active Comparator): NBI-6024 0.1 mg
  Interventions: Drug: NBI-6024
- 2 Experimental (Active Comparator): NBI-6024 0.5 mg
  Interventions: Drug: NBI-6024
- 3 Experimental (Active Comparator): NBI-6024 1 mg
  Interventions: Drug: NBI-6024
- 4 placebo (No Intervention): Placebo injection

INTERVENTIONS:
Drug: NBI-6024 — 0.1, 0.5 or 1 mg NBI-6024 First 3 doses every 2 weeks. Remaining doses given monthly. Total duration of dosing 24 months. Placebo controlled.
  Arms: 1 Experimental; 2 Experimental; 3 Experimental

SUMMARY:
This was a study designed to evaluate the efficacy of multiple doses of an investigational drug, NBI-6024, in adult (18 to 35 years of age) and adolescent (10 to 17 years of age) patients with new onset type 1 diabetes mellitus, on endogenous insulin production.

A total of 188 patients were enrolled in the study. The study was divided into three periods: screening, treatment (comprising an induction phase and maintenance phase), and follow-up.

NBI-6024 was generally well tolerated and exhibits a benign safety profile, as there were no significant safety issues with NBI-6024 treatment. In summary, NBI-6024 did not demonstrate statistically significant efficacy compared with placebo.

DETAILED DESCRIPTION:
This was a Phase II, multicenter (international), randomized, double-blind, placebo-controlled, parallel, dose-ranging study to evaluate the efficacy of multiple doses of an altered peptide ligand, NBI-6024, in adult (18 to 35 years of age) and adolescent (10 to 17 years of age) patients with new onset type 1 diabetes mellitus.

Study drug was administered subcutaneously a total of 26 times over a 24-month period. The first three doses were administered every 2 weeks (induction phase); all subsequent dosing occurred monthly (maintenance phase). Patients returned to the study center to receive study drug and have efficacy and safety assessments collected. The primary efficacy endpoint was the 2-hour peak C-peptide at Month 24. Other secondary analyses included AUC C-peptide, prescribed insulin usage, AUC blood glucose, HbA1c, hypoglycemic events, and hyperglycemic events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the age of 12 and 35 years, inclusive (changed to between the age of 10 and 35 years, inclusive, under Amendment 2)
* If female of childbearing potential, patient must use an acceptable method of birth control prior to and for 30 days post study
* Adult (greater than or equal to 18 years) female patients who were not of childbearing potential must be 2 years postmenopausal, or have had a hysterectomy or tubal ligation
* Were newly diagnosed with type 1 diabetes mellitus
* Presence of one or more of the following:

  * Anti-ICA512 antibodies
  * Anti-GAD antibodies
  * Anti-insulin antibodies, provided that the patient was not on insulin therapy for greater than 1 week
* Body mass index (BMI) < 28 kg/m2
* Stimulated serum C-peptide peak level between 0.4 pmol/mL and 3.0 pmol/mL, inclusive, at the time of screening
* Laboratory and 12-lead electrocardiogram (ECG) results within normal ranges or, if abnormal, considered by the investigator as non clinically significant for the safety and well being of the patient or for the purposes of the study

Exclusion Criteria:

* Use of an excluded medication/therapy including any of the following:

  * Steroids
  * Oral hypoglycemic agents
  * Chemotherapy and radiation
  * Immunosupressants
  * Nicotinamide >100 mg per day
  * Any drugs containing sibutramine
* Female patients with a positive pregnancy test or who are lactating
* Adult patients with body weight <45 kg; adolescent patients with body weight <30 kg; 10- and 11-year-old patients with body weight <25 kg
* History of cancer or have existing or actively managed cancer
* History of severe or anaphylactic allergic reactions
* Patients suffering from active skin infections that would prevent subcutaneous injection
* Positive test for HIV antigens, hepatitis B surface antigen, or hepatitis C antibodies
* History of alcohol or substance abuse

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 188 (Actual)
Dates: Start 2001-12; Primary Completion 2006-04 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To assess the effect of repeated administrations of NBI-6024 on endogenous insulin production as measured by C-peptide levels in adult and adolescent patients with new onset type 1 diabetes mellitus | monthly assessments, up to 24 months (end of study)

SECONDARY OUTCOMES:
To examine the effects of repeated administrations of NBI-6024 on insulin usage, glycemic control, and immune function (immunodynamics and pharmacodynamics) To examine the safety and tolerability of repeated administrations of NBI-6024 | monthly assessments, up to 24 months (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Areti Philotheou, MD, Principal Investigator — New Groote Schuur Hospital, Capetown, South Africa
Locations (21):
- Canada (3):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Center Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre de recherche clinique de Laval, Laval
- Czechia (2):
  - University Hospital and School of Medicine, Olomouc
  - Faculty Hospital Motol, Prague
- Helsinki University Hospital, Helsinki, Finland
- France (2):
  - Hôpital Debrousse, Lyon
  - Hôpital St Vincent de Paul, Paris
- Germany (2):
  - Diabetes Center for Children and Adolescents, Hanover
  - Institut für Diabetesforschung, München
- South Africa (6):
  - New Groote Schuur Hospital, Cape Town
  - Parklands Medical Center, Durban
  - Center for Diabetes and Endocrinology, Johannesburg
  - Donald Gordon Medical Center, Johannesburg
  - Medigate Medical Center, KwaZulu Natal
  - Helderberg Diabetic Clinic and Practice, Somerset West
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de Cruces, Cruces-Baracado
  - Hospital Materno-Infantil, Málaga
  - University Hospital Virgen del Rocío, Seville
- Maternal and Child Health Services 2, Dundee, United Kingdom

REFERENCES:
- [Derived] Walter M, Philotheou A, Bonnici F, Ziegler AG, Jimenez R; NBI-6024 Study Group. No effect of the altered peptide ligand NBI-6024 on beta-cell residual function and insulin needs in new-onset type 1 diabetes. Diabetes Care. 2009 Nov;32(11):2036-40. doi: 10.2337/dc09-0449. Epub 2009 Aug 18. PMID 19690081